CLINICAL TRIAL: NCT00342082
Title: A Pilot Study to Investigate Micronucleated Erythrocyte Frequencies in Infants Exposed to Nucleoside Antiretrovial Drugs in Utero and for 6 Weeks Postnatally
Brief Title: Effects of Anti-HIV Therapy on Red Blood Cells of HIV-infected Mothers and Their Infants
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904242; 04-E-N242
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-12-28

CONDITIONS: Cord Blood
Keywords: Zidovudine; HIV; Cord Blood

SUMMARY:
This collaborative investigation between NIEHS, Duke University, and the University of North Carolina (UNC) will study red blood cells of babies born to HIV-infected women receiving anti-retroviral treatment. Studies have shown that newborn mice whose mothers were given anti-HIV medications during pregnancy had abnormal red blood cells circulating in their blood stream, indicating genetic damage to the cells caused by the anti-HIV medications. It is not known if similar red blood cell abnormalities develop in human infants whose mothers received anti-HIV medication during their pregnancy. This study will examine red blood cells from infants exposed to anti-HIV medications and from non-exposed infants to look for differences between them involving this specific genetic damage.

Healthy pregnant women and HIV-infected pregnant women who received antiretroviral treatment during their last trimester of pregnancy and during labor may be eligible for this study. Babies of HIV-infected women are also included in the study. Candidates will be recruited from medical centers at Duke University and the UNC. HIV-infected mothers must plan to have their baby followed by either the UNC or the Duke Pediatric Infectious Disease clinic.

All women in the study will have 1 milliliter (less than 1/2 teaspoon) of blood collected for this study during delivery at the same time that other blood samples are obtained for their medical care. In addition, 5 ml (1 teaspoon) of umbilical cord blood will also be collected for this study at the time of delivery after the cord is no longer attached to the baby. This concludes participation of non-HIV infected women.

Babies born to HIV-infected mothers will have 1 ml of blood drawn between 0 to 3 days of life, between 4 to 6 weeks of life, and between 4 to 6 months of life. These bloodsamples will be collected at the same time as other routine scheduled blood draws.

DETAILED DESCRIPTION:
This is an observational study of pregnant women and their newborns. The population will include 10 HIV infected women on any antiretroviral regimen and their newborn infants and 10 healthy women on no antiretroviral regimen and their newborn infants.

Primary Objective: To determine if micronucleated erythrocytes can be detected more frequently in cord blood of infants exposed to zidovudine in utero and intrapartum compared to cord blood from infants not exposed.

Secondary Objectives:

* To determine if micronucleated erythrocytes can be detected in pregnant women on any antiretrovial agents.
* To determine if micronucleated erythrocytes change in frequency in infants exposed to antiretrovial agents over the first 6 weeks of life, during the time the infant is exposed to Zidovudine.
* To determine the change in micronucleated erythrocytes in the infants after cessation or Zidovudine (6 months).

ELIGIBILITY:
* INCLUSION CRITERIA: (Treated Group)
* HIV-infected
* Pregnant
* Treatment with antiretroviral regimen

INCLUSION CRITERIA: (Control Group)

-Healthy Pregnant Female

EXCLUSION CRITERIA: (Treated Group)

-None

EXCLUSION CRITERIA: (Control Group)

-Delivery less than 32 weeks gestation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0
Dates: Start 2004-06-25; Study Completion 2007-12-28

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - NIEHS, Research Triangle Park, Research Triangle Park, North Carolina

REFERENCES:
- [Background] Connor EM, Sperling RS, Gelber R, Kiselev P, Scott G, O'Sullivan MJ, VanDyke R, Bey M, Shearer W, Jacobson RL, et al. Reduction of maternal-infant transmission of human immunodeficiency virus type 1 with zidovudine treatment. Pediatric AIDS Clinical Trials Group Protocol 076 Study Group. N Engl J Med. 1994 Nov 3;331(18):1173-80. doi: 10.1056/NEJM199411033311801. PMID 7935654